CLINICAL TRIAL: NCT01556230
Title: Prospective Study of Clinically Nonfunctioning Pituitary Adenomas
Acronym: PAPS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine, Columbia University
Other Study IDs: AAAE1260; R01NS070600 (NIH)
Record Dates: First submitted 2012-03-09; First posted 2012-03-16 (Estimated); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pituitary Adenoma; Pituitary Tumor
Keywords: pituitary gland; pituitary adenoma; pituitary tumor; hypophysis; endocrine; neuroendocrine; hormone
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Serum and Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: The first group of subjects, Group I, will be followed in Protocol I and are a group of subjects with an apparent clinically nonfunctioning pituitary lesion who will be studied in a prospective study of conservative non-surgical management.
- Group II: A second group of subjects, Group II, are subjects who are undergoing surgical intervention for CNFA or radiotherapy for CNFA and these subjects will be studied in a prospectively follow up as part of Protocol II.
  Interventions: Procedure: Surgical intervention for CNFA; Radiation: Radiotherapy for CNFA

INTERVENTIONS:
Procedure: Surgical intervention for CNFA — (non-experimental) standard procedure
  Groups: Group II
Radiation: Radiotherapy for CNFA — (non-experimental) standard procedure
  Groups: Group II

SUMMARY:
This project is the first comprehensive prospective study of clinically non-functioning pituitary adenomas (CNFAs). Two groups of subjects will be studied: Group I will consist of 100 patients with clinically non-functioning (CNF) pituitary lesions who are asymptomatic and do not require surgery; Group II will consist of 250 patients who have pituitary lesions that are symptomatic and require surgery. Patients will be followed with a series of endocrine laboratory testing, physical examinations, testing of quality of life and neurocognitive function before and serially over time either during non-surgical management or after surgery and in some patients before and after radiotherapy (RT). Data on pituitary magnetic resonance imaging (MRI) studies and visual field testing being done over time during follow up as part of clinical care will be collected.

DETAILED DESCRIPTION:
PROTOCOL I: Prospective Study of the outcome of conservative non-surgical management of patients with asymptomatic, clinically non-functioning (CNF) pituitary lesions. This protocol will evaluate prospectively the outcome of non-surgical management of clinically non-functioning pituitary lesions that do not appear to need surgery as their initial therapy. The overall design consists of an initial baseline evaluation and then serial prospective follow up studies over time for up to 5 years of follow up. The study will evaluate laboratory testing, clinical examinations, quality of life and neurocognitive function in these patients. Data will be collected on visual fields and MRI studies of the pituitary tumor that are done prospectively as part of clinical care to evaluate these patients.

PROTOCOL II : Prospective study of the outcome of patients with symptomatic, clinically non-functioning pituitary tumors who are treated with transsphenoidal surgery and in some cases also radiotherapy. This protocol will evaluate prospectively the outcome of surgical management of asymptomatic clinically nonfunctioning pituitary lesions. The overall design consists of an initial baseline evaluation and then serial prospective follow up studies over time with up to 5 years of follow up. The study will evaluate laboratory testing, clinical examinations, quality of life and neurocognitive function in these patients. Data will also be collected on visual fields and MRI studies of the pituitary tumor that are done prospectively as part of clinical care to evaluate these patients. Data will be analyzed to determine the safety of observation alone following surgery for patients who do not have a clinically significant tumor remnant, if the silent corticotroph tumor type is characterized by elevated plasma levels of ACTH or its precursor, POMC, and if it is associated with an increased tumor recurrence rate. A group of patients who are planning RT will also be studied by these same procedures before and after RT in order to determine if the outcomes of patients who receive RT for treatment of tumor re-growth to that of those who do not receive RT with respect to further tumor growth, endocrine or neurological dysfunction. Quality of life and neurocognitive function in patients with clinically non-functioning pituitary lesions treated with surgery alone or those who also receive radiotherapy will be prospectively assessed.

ELIGIBILITY:
GROUP I

Inclusion Criteria:

* adult patients with pituitary lesions that do not require surgical intervention.
* pituitary lesion that has been demonstrated on a magnetic resonance imaging (MRI) to be consistent with an adenoma (not a cystic lesion such as a Rathke's cleft cyst).
* patients with macroadenomas (> 1 cm) or large microadenomas 6-9 mm.
* a prolactin level < 40 ng/ml.

Exclusion Criteria:

* presence of visual or neurological deficits due to the tumor, tumor impingement on the optic chiasm and physical or laboratory abnormalities consistent with a biologically active hormone secreting tumor.

GROUP II

Inclusion Criteria:

* adult patients with pituitary lesions that require surgical intervention and are planning on surgery or who had surgery in the past and are now undergoing pituitary radiotherapy.
* pre-surgery patients will have a pituitary lesion that has been demonstrated on a MRI to be consistent with an adenoma (not a cystic lesion such as a Rathke's cleft cyst) and that is a macroadenoma (> 1 cm).
* presence of visual or neurological deficits due to the tumor or impingement of the tumor on the optic chiasm is permitted.
* a prolactin level < 100 ng/ml if lesion is > or = 10 mm in size or a prolactin level < 40 ng/ml if lesion is < 10 mm in size.
* patients with mild/moderate hyperprolactinemia and recommended for dopamine agonist therapy (on the chance that the lesion is truly a prolactinoma) may re-enter the study should they be a dopamine agonist failure and require surgery.
* patients with hypopituitarism and no other surgical indication that choose to undergo surgery is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any persons diagnosed with a non-functioning pituitary adenoma that is willing to travel to our study center at Columbia University in New York for all study visits.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2024-06 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with pituitary tumor enlargement | 5 years
  Tumor enlargement over the study period

SECONDARY OUTCOMES:
Change in neurocognitive function test score | Baseline, 5 years
  Neurocognitive function change over the time frame of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U. Freda, MD, Principal Investigator — Columbia University College of Physicians&Surgeons
Locations (1):
- Columbia University Vagelos College of Physicians & Surgeons, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided